CLINICAL TRIAL: NCT05743309
Title: Evaluation of Telemedicine Practices for Contraceptive Counseling Given to Pregnant Women During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Evaluation of Telemedicine Practices for Contraceptive Counseling During the COVID-19 Pandemic: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rabia Saglam Aksut, Asst. Prof., Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FenerbahçeU
Record Dates: First submitted 2023-02-22; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Family Planning Services; Telemedicine; Pregnant Women; Women's Health; COVID-19 Pandemic
Keywords: Family Planning Services; Telemedicine; Pregnant Women; Women's Health; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In this study, there are two groups (one experimental and one control group). While experimental group patients received telemedicine practices related to Family planning, control group patients received only routine health services provided by primary health care setting.
Who Masked: Participant
Masking Description: Participants did not know which group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Practices (Experimental): In this study, telemedicine practices stand for video call sessions used for contraceptive counseling services.
  Interventions: Behavioral: Video call sessions
- Routine Contraceptive Counseling Services (No Intervention): Participants in the control group received only routine contraceptive counseling services provided by primary health care settings.

INTERVENTIONS:
Behavioral: Video call sessions — Investigators made video call sessions with the participants.
  Arms: Telemedicine Practices

SUMMARY:
The goal of this randomized clinical trial is to evaluate the telemedicine practices for contraceptive counseling given to pregnant women during the COVID-19 pandemic. The main questions it aims to answer are:

* Does family planning counseling given to pregnant women by using telemedicine practices have an effect on the knowledge level about family planning?
* Is family planning counseling given to pregnant women by using telemedicine practices effective on satisfaction with family planning services? Participants have attended to contraceptive counseling video call sessions provided via WhatsApp application and they have the opportunity to see the consultant and her materials during these sessions. After these sessions (two weeks later), contraceptive counseling video call session has been repeated, and at the end of this second session, women have been asked to answer the questions in the "Family Planning Knowledge Level Form" and the "Family Planning Services Satisfaction Scale". There is a comparison group (a control group) in this study, and no intervention was made to the women in the control group other than the routine services given in primary care settings.

Researchers will compare the experimental group with control group to see if the telemedicine practices are effective in increasing the knowledge level of pregnant women about family planning and in the satisfaction of family planning services provided by primary health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Women in the third trimester of their pregnancy and who agreed to participate in the study have been included in this study.

Exclusion Criteria:

* Women with psychiatric disorder have been excluded from this study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Family planning counseling given to pregnant women by using telemedicine practices have an effect on the knowledge level about family planning and on the satisfaction with family planning services. | 6 Months
  Primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahce University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steenland MW, Geiger CK, Chen L, Rokicki S, Gourevitch RA, Sinaiko AD, Cohen JL. Declines in contraceptive visits in the United States during the COVID-19 pandemic. Contraception. 2021 Dec;104(6):593-599. doi: 10.1016/j.contraception.2021.08.003. Epub 2021 Aug 14. PMID 34400152
- [Result] Stifani BM, Avila K, Levi EE. Telemedicine for contraceptive counseling: An exploratory survey of US family planning providers following rapid adoption of services during the COVID-19 pandemic. Contraception. 2021 Mar;103(3):157-162. doi: 10.1016/j.contraception.2020.11.006. Epub 2020 Nov 17. PMID 33212033
- [Result] Martinez KA, Rastogi R, Lipold L, Rothberg MB. Response to requests for contraception in one direct-to-consumer telemedicine service. Contraception. 2020 May;101(5):350-352. doi: 10.1016/j.contraception.2020.01.017. Epub 2020 Feb 12. PMID 32059840
- [Result] Stifani BM, Madden T, Micks E, Moayedi G, Tarleton J, Benson LS. Society of Family Planning Clinical Recommendations: Contraceptive Care in the Context of Pandemic Response. Contraception. 2022 Sep;113:1-12. doi: 10.1016/j.contraception.2022.05.006. Epub 2022 May 18. PMID 35594989
- [Result] Huang I, Delay R, Boulware A, McHugh A, Wong ZJ, Whitaker AK, Stulberg D, Hasselbacher L. Telehealth for contraceptive care: Lessons from staff and clinicians for improving implementation and sustainability in Illinois. Contracept X. 2022 Aug 14;4:100083. doi: 10.1016/j.conx.2022.100083. eCollection 2022. PMID 36060498
- [Result] Stifani BM, Smith A, Avila K, Boos EW, Ng J, Levi EE, Benfield NC. Telemedicine for contraceptive counseling: Patient experiences during the early phase of the COVID-19 pandemic in New York City. Contraception. 2021 Sep;104(3):254-261. doi: 10.1016/j.contraception.2021.04.006. Epub 2021 Apr 20. PMID 33861981
- [Result] Mickler AK, Carrasco MA, Raney L, Sharma V, May AV, Greaney J. Applications of the High Impact Practices in Family Planning during COVID-19. Sex Reprod Health Matters. 2021 Dec;29(1):1881210. doi: 10.1080/26410397.2021.1881210. PMID 33599196
- [Result] Karaahmet AY, Bilgic FS. COVID-19: the unmet need for family planning and its effects on sexuality: a cross-sectional study. Rev Assoc Med Bras (1992). 2022 Jun 24;68(6):827-832. doi: 10.1590/1806-9282.20220138. eCollection 2022. PMID 35766699
- [Result] Miller HE, Henkel A, Leonard SA, Miller SE, Tran L, Bianco K, Shaw KA. The impact of the COVID-19 pandemic on postpartum contraception planning. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100412. doi: 10.1016/j.ajogmf.2021.100412. Epub 2021 May 28. PMID 34058421
- [Result] Sileo KM, Muhumuza C, Helal T, Olfers A, Lule H, Sekamatte S, Kershaw TS, Wanyenze RK, Kiene SM. Exploring the effects of COVID-19 on family planning: results from a qualitative study in rural Uganda following COVID-19 lockdown. Reprod Health. 2023 Feb 9;20(1):31. doi: 10.1186/s12978-023-01566-3. PMID 36759838
- [Result] Krishna UR. Reproductive Health During the COVID-19 Pandemic. J Obstet Gynaecol India. 2021 Aug;71(Suppl 1):7-11. doi: 10.1007/s13224-021-01546-2. Epub 2021 Aug 30. PMID 34483512